CLINICAL TRIAL: NCT03004768
Title: Pharmacokinetics and Metabolism of [14C]BMS-986165 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-016
Record Dates: First submitted 2016-12-19; First posted 2016-12-29 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose of radiolabeled BMS-986165 (Experimental)
  Interventions: Drug: BMS-986165

INTERVENTIONS:
Drug: BMS-986165 — Oral solution dose of 24 mg [14C] BMS-986165 containing approximately 100 micro Ci of TRA

SUMMARY:
An oral dose in healthy subjects to obtain information about the absorption, metabolism, and excretion (AME) of BMS-986165

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Target population: Healthy males with no clinically significant deviations from normal in medical history, physical examinations, vital signs, electrocardiograms (ECGs), physical measurements, and clinical laboratory tests
* Body weight of at least 50 kilograms (110 pounds); body mass index (BMI) between 18 to 32 kg/m2.
* No evidence of acute infection or other significant problem as determined from a review of a chest x-ray, medical history, and physical examination

Exclusion Criteria:

* History of any chronic or acute illness including active TB in the last 3 years, recent infection, gastrointestinal disease, smoking within less than 6 months prior to dosing, alcohol abuse, inability to tolerate oral medication, or inability to be venipunctured.
* Vaccination or plans for vaccination with any live vaccine 12 weeks prior to first dose of study drug, during the course of the study
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, electrocardiograms, or clinical laboratory determinations beyond what is consistent with the target population.
* Participant with greater than Grade 2 acne.
* Participated in a radiolabeled drug study within the previous 12 months; clinically significant diagnostic or therapeutic radiation exposure within the previous 12 months; or current employment in a job requiring radiation exposure monitoring.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is PK exposure that will be determined from plasma concentration versus time | Day 1 to Day 13
Urinary/fecal TRA (Total radioactivity) recovery data | Day 1 to Day 13
PK terminal elimination half-life data (T-HALF) | Day 1 to Day 13
PK apparent total body clearance (CL/F) | Day 1 to Day 13
PK apparent volume of distribution (Vz/F) | Day 1 to Day 13
PK time of maximum observed plasma concentration (Tmax) | Day 1 to Day 13

SECONDARY OUTCOMES:
Safety endpoints include the incidence of adverse events (AEs) | Day 1 to Day 13
Safety endpoints include the results of electrocardiogram tests (ECGs) | Day 1 to Day 13
Safety endpoints include the results of vital signs | Day 1 to Day 13
Safety endpoints include the results of physical exams | Day 1 to Day 13
Safety endpoints include the results of clinical laboratory tests | Day 1 to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Madison Clinical Research Unit, Madison, Wisconsin, United States

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/